CLINICAL TRIAL: NCT06829628
Title: The Effects of Teaching Strategies Integrating a Mobile Chatbot with ARCS-V Motivation Theory on Learning Motivation and Performance in Medical-Surgical Nursing
Brief Title: A Mobile Chatbot with ARCS-V Motivation Theory on Learning Motivation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Miao-Yi Chen, Investigator, Chang Gung University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CGUST Chiayi campus
Record Dates: First submitted 2025-02-08; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Nursing Education Research; Chatbot-Based Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Nursing students receiving chatbot-based learning.
  Interventions: Behavioral: chatbot teaching strategies
- Control Group (No Intervention): No Intervention

INTERVENTIONS:
Behavioral: chatbot teaching strategies — Chatbot-Based Learning
  Arms: Intervention Group

SUMMARY:
This study will implement a smartphone chatbot in medical-surgical nursing education to enhance nursing students' learning motivation and academic performance. T

ELIGIBILITY:
Inclusion Criteria:

* Second-year Nursing students
* Taking an adult nursing course
* Aged 18 or older
* Willing to voluntarily participate in this study

Exclusion Criteria:

* Students auditing the course

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-17 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
learning motivation | Baseline, 9 weeks, and 18 weeks after intervention
  The Course Interest Survey will be used to measure learning motivation. It consists of 34 items, with responses rated on a 5-point scale, where 1 indicates "Not true" (completely not applicable) and 5 indicates "Very true" (completely applicable). Higher scores indicate greater learning motivation.

IPD SHARING:
Plan to Share IPD: No